CLINICAL TRIAL: NCT02020785
Title: Randomized Cross-over Study Examining the Effects of Phosphorus Additives on Urinary Albumin Excretion and Fibroblast Growth Factor-23
Brief Title: Study of Dietary Additive Phosphorus on Proteinuria and Fibroblast Growth Factor-23
Acronym: SODA-POP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Alexander Chang, Clinical Investigator, Geisinger Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00082089; 13CRP16970085 (Other Grant/Funding Number: American Heart Association); Satellite Dialysis (Other Grant/Funding Number: National Kidney Foundation)
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Albuminuria
Keywords: proteinuria
MeSH Terms: conditions — Albuminuria; Proteinuria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher phosphorus period (Active Comparator): Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  Interventions: Other: Higher phosphorus period
- Lower phosphorus period (Placebo Comparator): Commercially-available unaltered food/beverage products without phosphorus additives (<10mg/d of phosphorus) will be given for 3 weeks
  Interventions: Other: Lower phosphorus period

INTERVENTIONS:
Other: Higher phosphorus period — Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks.
  All participants at the beginning of the study will receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives.
  Arms: Higher phosphorus period
Other: Lower phosphorus period — Commercially-available unaltered food/beverage products without phosphorus additives (<10mg/d of phosphorus) will be given for 3 weeks.
  All participants at the beginning of the study will receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives.
  Arms: Lower phosphorus period

SUMMARY:
Phosphorus-based food additives are commonly used by food manufacturers for many applications, such as enhancing flavor, in ready-to-eat foods and beverages. While these additives can significantly increase an individual's daily phosphorus intake, little is known about the effect of dietary phosphorus on kidney health. In this study, the investigators will first lower baseline phosphorus intake to about 1000mg/d by educating participants to avoid foods with phosphorus additives. Then, participants will be randomized to a higher phosphorus period (~2gm/d) and a lower phosphorus period (~1gm/d) by providing unaltered, commercially-available food/beverage products with and without phosphorus additives.

The investigators hypothesize that participants will have higher urine albumin excretion and fibroblast growth factor-23 (FGF-23) during the higher phosphorus period compared to the lower phosphorus period.

DETAILED DESCRIPTION:
The Study of Dietary Additive Phosphorus on Proteinuria and FGF-23 (SODA-POP) was a single-center, randomized, double-blind, two-period cross-over study that examined the effect of higher vs. lower phosphorus intake for 3 week periods, achieved by addition of commercially available diet beverages and breakfast bars to diet on albuminuria and fibroblast growth factor 23, in adults with presumed early chronic kidney disease (estimated glomerular filtration rate >= 45 ml/min/1.73m2; and urine albumin/creatinine ratio >=17 mg/g for men or >=25 mg/g for women).

ELIGIBILITY:
Inclusion Criteria:

Adults at least 21 years of age with at least microalbuminuria

Exclusion Criteria:

Estimated glomerular filtration rate <45ml/min/1.73m2, poorly controlled diabetes or hypertension, nephrotic syndrome, hyperparathyroidism, Paget's Disease, multiple myeloma, uncontrolled thyroid disease, chronic antacid use, use of phosphorus binders, phosphorus supplements, or high-dose vitamin D, inability to complete feeding study, investigator discretion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Chang, MD, MS, Principal Investigator — Geisinger Clinic; Lawrence J Appel, MD, MPH, Study Director — Johns Hopkins University
Locations (1):
- Prohealth Clinical Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Chang A, Batch BC, McGuire HL, Vollmer WM, Svetkey LP, Tyson CC, Sanguankeo A, Anderson C, Houston J, Appel LJ. Association of a reduction in central obesity and phosphorus intake with changes in urinary albumin excretion: the PREMIER study. Am J Kidney Dis. 2013 Nov;62(5):900-7. doi: 10.1053/j.ajkd.2013.04.022. Epub 2013 Jun 28. PMID 23810691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary recruitment strategies included mass mailing of study brochures to individuals with self-reported type 2 diabetes in neighboring zip codes and to past and current participants of other research studies.
Groups:
- Higher Phosphorus Period First, Then Lower Phosphorus Period: Randomized to higher phosphorus period first, then lower phosphorus period second.
  Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  At the beginning of the study participants receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives
  Higher phosphorus period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
  Lower phosphorus period: Commercially-available unaltered food/beverage products without any phosphorus additives given for 3 weeks
- Lower Phosphorus Period First, Then Higher Phosphorus Period: Randomized to higher phosphorus period first, then lower phosphorus period second.
  Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  At the beginning of the study participants receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives
  Lower phosphorus period: Commercially-available unaltered food/beverage products without any phosphorus additives given for 3 weeks
  Higher phosphorus period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
Period: First Intervention (3 Weeks)
Arm/Group | Higher Phosphorus Period First, Then Lower Phosphorus Period | Lower Phosphorus Period First, Then Higher Phosphorus Period
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Higher Phosphorus Period First, Then Lower Phosphorus Period | Lower Phosphorus Period First, Then Higher Phosphorus Period
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Higher Phosphorus Period Then Lower Phosphorus Period: Randomized to higher phosphorus period first, then lower phosphorus period second.
  Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  At the beginning of the study participants receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives
  Higher phosphorus period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
  Lower phosphorus period: Commercially-available unaltered food/beverage products without any phosphorus additives given for 3 weeks
- Lower Phosphorus Period Then Higher Phosphorus Period: Randomized to higher phosphorus period first, then lower phosphorus period second.
  Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  At the beginning of the study participants receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives
  Lower phosphorus period: Commercially-available unaltered food/beverage products without any phosphorus additives given for 3 weeks
  Higher phosphorus period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
- Total: Total of all reporting groups
Arm/Group | Higher Phosphorus Period Then Lower Phosphorus Period | Lower Phosphorus Period Then Higher Phosphorus Period | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (7.3) | 64.2 (9.9) | 66.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 16 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 14 | 28
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Urine Albumin Excretion
Description: Two 24-hour urine collections will be collected during the 3rd week of each period
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: mg/day
Groups:
- Higher Phosphorus Period; Lower Phosphorus Period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) will be given for 3 weeks
  At the beginning of the study participants receive dietary education to reduce their baseline consumption of phosphorus to a goal of ~1gm/d by receiving education on avoiding phosphorus-based additives.
  Patients then randomized to higher phosphorus period or lower phosphorus period first.
  Higher phosphorus period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
  Lower phosphorus period: Commercially-available unaltered food/beverage products without any phosphorus additives given for 3 weeks
Arm/Group | Higher Phosphorus Period | Lower Phosphorus Period
Number analyzed (Participants) | 31 | 31
mg/day | 86.2 [51.8 to 143.4] | 76.4 [47.2 to 123.8]
Statistical Analysis 1: Comparison: Higher Phosphorus Period vs Lower Phosphorus Period; Sample size for this study was calculated using the xsampsi module in STATA, based on a previous study with repeat 24-hour urine collections (standard deviation, 1.04). At an α level of 0.05, we anticipated that a sample size of 30 participants with mean albuminuria of 100 mg/d would result in >80% power to detect a 13% difference in log- transformed albuminuria between the higher and lower phosphorus additive periods; Test type: Superiority — Main analyses were intention-to-treat using mixed effects models allowing intercepts to vary for each individual. Carryover effects were examined by using treatment by assignment-order interaction terms. Pre-specified sensitivity analyses were conducted excluding patients who were non-compliant, prior to data analysis: 1st, noncompliance based on missing product pickups and follow-up visits; 2nd, suspected poor compliance (< 250 mg difference between the higher and lower period).]; p = 0.05, Mixed Models Analysis — For each outcome, a p value < 0.05 was considered statistically significant without adjustment for multiple comparisons; Mean Difference (Final Values) = 0.143, 95% CI 2-sided [-0.025 to 0.34] — Estimate (14.3%, 95% CI: -2.5%, 34.0%) is the estimated difference between end of higher phosphorus period and end of lower phosphorus period from mixed effects analyses for log-transformed 24-hour urine albumin excretion

2. Primary Outcome: Fibroblast Growth Factor-23 (FGF-23)
Description: Plasma FGF-23 will be measured at the end of each 3 week period in the morning after an overnight fast.
  As this is a small pilot study, we will not adjust for multiple comparisons. A p value<0.05 will be considered statistically significant for both outcomes
Time Frame: 3 weeks
Measure: Geometric Mean (95% Confidence Interval); unit: Relative units/ml
Arm/Group | Higher Phosphorus Period | Lower Phosphorus Period
Number analyzed (Participants) | 31 | 31
Relative units/ml | 132.6 [115.4 to 152.3] | 128.2 [113.1 to 145.3]
Statistical Analysis 1: Comparison: Higher Phosphorus Period vs Lower Phosphorus Period; Test type: Superiority; p = 0.05, Mixed Models Analysis — For each outcome, a p value < 0.05 was considered statistically significant without adjustment for multiple comparisons; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [-0.059 to 0.136] — Estimate (3.4%, 95% CI: -5.9%, 13.6%) is the estimated difference between end of higher phosphorus period and end of lower phosphorus period from mixed effects analyses for log-transformed fibroblast growth factor 23

3. Secondary Outcome: Systolic Blood Pressure
Description: Blood pressure was measured at the end of weeks 1, 2, and 3. At each visit, 3 readings were obtained in the seated position by trained and certified observers after 5 minutes of rest with an Omron HEM-907 device (Omron Healthcare Inc, Bannockburn, Ill) using a standardized protocol. We used the average of all blood pressure measurements at the end of weeks 1, 2, and 3 for each period.
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Higher Phosphorus Period | Lower Phosphorus Period
Number analyzed (Participants) | 31 | 31
mmHg | 126.9 (13.5) | 128 (15.6)
Statistical Analysis 1: Comparison: Higher Phosphorus Period vs Lower Phosphorus Period; Test type: Superiority; p = 0.05, Mixed Models Analysis — For each outcome, a p value < 0.05 was considered statistically significant without adjustment for multiple comparisons; mean difference (during each period) = -1.1, 95% CI 2-sided [-4.1 to 1.9]

4. Secondary Outcome: Diastolic Blood Pressure
Description: Blood pressure measured at the end of weeks 1, 2, and 3. At each visit, 3 readings were obtained in the seated position by trained and certified observers after 5 minutes of rest with an Omron HEM-907 device (Omron Healthcare Inc, Bannockburn, Ill) using a standardized protocol. We used the average of all these readings taken during end of weeks 1, 2, and 3 for each period.
Time Frame: 2-3 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Higher Phosphorus Period | Lower Phosphorus Period
Number analyzed (Participants) | 31 | 31
mmHg | 69.3 (10.8) | 70.2 (11.4)
Statistical Analysis 1: Comparison: Higher Phosphorus Period vs Lower Phosphorus Period; Test type: Superiority; p = 0.05, Mixed Models Analysis — For each outcome, a p value < 0.05 was considered statistically significant without adjustment for multiple comparisons; mean difference (during each period) = -0.8, 95% CI 2-sided [-2.7 to 1.0]

ADVERSE EVENTS:
Time Frame: At the end of each 3 week study period.
Description: Participants were asked at the end of each study period if they experienced possible side effects.
Groups:
- Higher Phosphorus Period: Commercially-available unaltered food/beverage products containing phosphorus additives (~1gm/d of phosphorus) given for 3 weeks
- Lower Phosphorus Period: Commercially-available unaltered food/beverage products without phosphorus additives (<10mg/d of phosphorus) given for 3 weeks
Arm/Group | Higher Phosphorus Period | Lower Phosphorus Period
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 22/31 | 23/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Phosphorus Period (N=31) | Lower Phosphorus Period (N=31)
Gastrointestinal symptoms (Gastrointestinal disorders) | 19 (19) | 21 (21) — Participants were asked at the end of each study period if they experienced possible side effects. The specific adverse event terms cannot be separated due to the manner in which this was assessed.
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 12 (12)
Flu-like symptoms (Infections and infestations) | 1 (1) | 3 (3)
Fatigue (General disorders) | 7 (7) | 7 (7)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)

LIMITATIONS AND CAVEATS:
Small sample size, short duration of intervention, changes in background diet during the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No